CLINICAL TRIAL: NCT03534128
Title: Influence of Visual, Auditory and Combinated Cues on Virtual Spatial Navigation in Brain-injured Patients.
Brief Title: Combinated Cues and Virtual Spatial Navigation
Acronym: CombiVirtual
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Centre Ressources Francilien du Traumatisme Crânien (Other)
Collaborators: Fondation Paul Bennetot (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: CombiVirtual
Record Dates: First submitted 2018-04-09; First posted 2018-05-23 (Actual); Last update posted 2018-08-28 (Actual); Status verified 2018-08

CONDITIONS: Traumatic Brain Injury
Keywords: Traumatic Brain Injury; Spatial navigation; Virtual Reality; Cues
MeSH Terms: conditions — Brain Injuries, Traumatic; Spatial Navigation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Spatial navigation evaluation (Experimental)
  Interventions: Other: Evaluation of the effect of cues on virtual spatial navigation using a virtual district

INTERVENTIONS:
Other: Evaluation of the effect of cues on virtual spatial navigation using a virtual district — Evaluation of the effect of cues on virtual spatial navigation using a virtual district

SUMMARY:
Many patients suffer from a topographical disorientation after a traumatic brain injury. Virtual Reality settings allow us to develop navigational cues, in order to rehabilitate patients or to help them in daily life. Some visual and auditory cues have proved efficient in helping patients navigating in a virtual environment but when administered separately, they never enabled patients to obtain a similar navigation performance as healthy controls. Moreover, the effect of the combination between visual and auditory cues has never been studied before. The objective of the present study is to determine if the combination between visual and auditory cues improve spatial navigation and memory of patients with a traumatic brain injury.

Therefore, the investigators intend to include in this prospective randomized study 45 patients who have had a moderate or severe traumatic brain injury and 20 healthy controls. Participants will have to reproduce actively with a joystick three different paths including 6 intersections that they have previously seen on a computer screen. One path will be done without cues, one with visual or auditory cues, and one with combined cues (visual+auditory). The order of the paths will be randomized. Auditory cues consist of beeping sounds indicating the direction at each intersection. Visual cues consist of salient landmarks (red and blinking) positioning at each intersection.

The main judgment criterion will be the number of trajectory mistakes during the path reproduction (/6). The secondary judgment criteria will be : time of navigation, memory of the landmarks, the route and the survey of the virtual environment. The confirmation of the help given by the combined cues could further allow the patients to use them in rehabilitation or in real life using augmented reality.

DETAILED DESCRIPTION:
* Main objective of the study: to determine if the combination between visual and auditory cues improve spatial navigation and memory of patients with a traumatic brain injury (TBI).
* Secondary objective of the study: to determine if the number of patients (%) with no trajectory mistakes with combined cues differs significantly from the one of healthy controls.
* Investigation centers: 4 : Rehabilitation Unit of Raymond Poincaré Hospital (Garches, France); Rehabilitation Unit of the University Hospital of Bordeaux (France); Rehabilitation Unit of the University Hospital of Rennes (France); Rehabilitation center of Kerpape (France)
* Study description: prospective, clinical, randomized, controlled
* Inclusion criteria: for the patients: history of moderate or severe traumatic brain injury with no other previous neurological history; for the healthy controls: no neurological history.
* Exclusion criteria: deafness (more than 40 decibels at one ear); low non-corrected visual acuity; severe comprehension issues; severe behavioral issues (DSM IV definition); epileptic seizures during the 6 months preceding the inclusion in the present study, except the 14 days after the TBI; a non-stabilized acute disease; absence of social assurance; ongoing legal protection; age under 18; pregnancy and breast-feeding
* Procedure: 1) Selection of patients by the investigators in each center. Verification of the inclusion and the exclusion criteria, and delivery of the information note.

  2) Visit 1: At least 24 hours later, investigators will gather the written consent of the participants. Then, participants will have to reproduce actively with a joystick three different paths including 6 intersections that they have previously seen on a computer screen representing a virtual district. One path will be done without cues, one with visual or auditory cues, and one with combined cues (visual+auditory). The order of the paths will be randomized. Auditory cues consist on beeping sounds indicating the direction at each intersection. Visual cues consist on salient landmarks (red and blinking) positioning at each intersection. The virtual district used looks like a North-American medium-sized town. Duration: 1h30 maximum.

  3) A second visit will be organized less than 15 days after the Visit 1. It will consist of a classical neuropsychological evaluation, assessing global cognitive efficiency (using the Mini Mental State Examination), memory (using the Gröber and Buschke test and the Rey Figure), executive functions (using the Frontal Assessment Battery and the Stroop test), attentional functions (using the Zazzo test), visuo-spatial functions (using the Rotation Mental test, the Santa Barbara Questionnaire and a mental imagery test developed by Maurer and Descloux) and neglect (using a barrage test and the Catherine Bergego scale). Duration: 2 hours maximum.
* Duration of the study: 18 months
* Number of participants included (using a calculation for the number of participants): 45 patients with a traumatic brain injury, and 20 healthy controls
* Statistics: comparisons between conditions will be done using ANOVA tests, then 2-by-2 using t-tests (if normality is established; if not, Kruskall-Wallis tests and Wilcoxon tests will be used). Correlations (Pearson or Spearman tests) will be done between spatial navigation performances and neuropsychological results at pencil-and-paper tasks.
* Ethics: The consent of an Ethics Committee has been requested (pending). A clinician Research Associate will monitor the results. A meeting with the investigators of the 4 centers will be planned every 6 months.
* The Source data verification will be done by the Clinician Research Associate for each participant.
* Reporting for adverse effects: the possible adverse effects are fatigue, headache, cyber-sickness (the same effect that can occur during the use of a computer) and exceptionally epileptic seizure (risk limited by the shortness of the exposure with the computer; 8 minutes per path on average). If a severe adverse effect occurs, like an epileptic seizure, it will be immediately reported to the sponsor, and a formulary will be send to a specific cell (named "Cellule Vigilance de la Fédération de Recherche Clinique"). The participation of the subject to the study will be immediately stopped.
* Plan for missing data: the presence of missing data or lost participants has been taken into account in the calculation for the number of participants. The data will be analyzed in "intention-to-treat".

ELIGIBILITY:
Inclusion Criteria:

1/ For the patients:

* History of moderate or severe traumatic brain injury with no other previous neurological history 2/ For the healthy controls:
* No neurological history

Exclusion Criteria:

* Deafness (more than 40 decibels at one ear)
* Low non-corrected visual acuity
* Severe comprehension issues
* Severe behavioral issues (DSM IV definition)
* Epileptic seizures during the 6 months preceding the inclusion in the present study, except the 14 days after the TBI
* A non-stabilized acute disease
* Absence of social assurance
* Ongoing legal protection
* Age under 18
* Pregnancy and breast-feeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 45 (Estimated)
Dates: Start 2018-06-20 (Actual); Primary Completion 2019-12-31 (Estimated); Study Completion 2019-12-31 (Estimated)

PRIMARY OUTCOMES:
Number of trajectory mistakes | 1-8 minutes
  Number of trajectory mistakes during the reproduction of the path (/6)

SECONDARY OUTCOMES:
Time of navigation | 1-8 minutes
  Time of navigation during the reproduction of the path (in seconds)
Memory of landmarks | 1-5 minutes
  After navigation, spelling of the landmarks of the district and classification of these landmarks in a chronological order
Memory of the route | 1-5 minutes
  After navigation, participants will have the recognize from a photography the direction that they have taken at each intersection
Memory of survey | 1-5 minutes
  After navigation, participants will be asked to choose one drawing representing their path between 4 possibilities

CONTACTS AND LOCATIONS:
Overall Officials: Mélanie Cogné, MD, PhD, Principal Investigator — Raymond Poincaré Hospital
Locations (4):
- France (4):
  - University Hospital of Bordeaux (Pellegrin), Bordeaux, Aquitaine
  - Rehabilitation Unit of Kerpape, Kerbach, Brittany Region
  - University Hospital of Rennes (Pontchaillou), Rennes, Brittany Region
  - Rehabilitation Unit, Raymond Poincaré Hospital, Garches, Île-de-France Region

IPD SHARING:
Plan to Share IPD: No